CLINICAL TRIAL: NCT03059043
Title: Prospective, Multicenter,Randomized Clinical Investigation of A Viscoelastic-free Method for Implantable Collamer Lens (ICL) Implantation to Treat High Myopia: A Pilot Study
Brief Title: Safety and Efficacy Study of A Viscoelastic-free Method for Implantable Collamer Lens (ICL) Implantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, A-Yong Yu, Director of the Cataract Clinical Center, Wenzhou Medical University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 20170121
Record Dates: First submitted 2017-02-13; First posted 2017-02-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Myopia
Keywords: Phakic Intraocular Lenses; viscoelastic
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- viscoelastic-free system (Experimental): Eyes in this group will use viscoelastic-free implantation system during the surgery
  Interventions: Device: viscoelastic-free implantation system
- viscoelastic-assisted system (Active Comparator): Eyes in this group will utilize the standard viscoelastic-assisted Implantation system during the surgery
  Interventions: Device: standard viscoelastic-assisted Implantation system

INTERVENTIONS:
Device: viscoelastic-free implantation system — Viscoelastic-free implantation system use balanced salt solution irrigation during the implantation
  Arms: viscoelastic-free system
Device: standard viscoelastic-assisted Implantation system — This method utilize the viscoelastic agent to fill and maintain the anterior chamber during the implantation
  Arms: viscoelastic-assisted system

SUMMARY:
This study evaluates the safety and efficacy of a viscoelastic-free method for Implantable Collamer Lens(ICL) implantation to treat high myopia. The subjects undergo randomization of ICL implantation using the viscoelastic-free method on one eye and undergoing standard method on the other one. The post-operative data are collected for analysis.

DETAILED DESCRIPTION:
Implantable Collamer Lens(ICL) implantation has been proved to be an effective refractive option for surgical correction of high myopia. Currently, standard method utilizing the viscoelastic agent to fill and maintain the anterior chamber during the implantation, this requires an additional step to remove the viscoelastic agent at the end of the surgery and may cause the intraocular pressure spike in the early post-operative phase due to the incomplete removal of the viscoelastics. The new method is viscoelastic-free, which can be achieved by using balanced salt solution irrigation during the implantation.

This study is a prospective, randomized, paired-eye study to compare the safety and efficacy of the viscoelastic-free method with the standard method. Subjects enrolled in the study will be randomized to receive viscoelastic-free method on one eye and undergo standard method on the other one.The clinical outcomes of two groups will be assessed at several follow-ups: 2 hours, 1 day, 1 week, 1 month, 3 months and 6 months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Documented stable refraction for at least 1 year(within 0.5D)
* Best spectacle-corrected visual acuity (BCVA) of 20/40 or better
* Clear central cornea
* -0.5D to -18.0D of myopic refractive error
* Normal anterior chamber depth at least 2.8 mm to endothelium
* Endothelial cell density (ECD) more than 2000 cell/mm2
* Pupil diameter smaller than 7.0 mm under mesopic condition
* Discontinued 3 weeks for hard contact lens and 1 week for soft contact lens wear

Exclusion Criteria:

* Preexisting ocular diseases or conditions other than myopia, evidence of progressive or acute ocular disease
* Evidence of connective tissue disease or other systemic diseases that may confound the results of the study;
* Narrow angle of anterior chamber
* Pregnant, lactating, or planning to become pregnant during the course of the trial

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-11-16 (Actual); Primary Completion 2026-06-22 (Estimated); Study Completion 2026-06-22 (Estimated)

PRIMARY OUTCOMES:
Early Post-operative Intraocular Pressure | 2 hours after surgery
  Intraocular Pressure measured by non-contact tonometers

SECONDARY OUTCOMES:
Corrected Visual Acuity (UCVA) at Distance | baseline, 1 day, 1 week, 1 month, 3 months and 6 months after surgery
  Subjective refraction
Uncorrected Visual Acuity (UCVA) at Distance | baseline, 1 day, 1 week, 1 month, 3 months and 6 months after surgery
  Measure by visual acuity chart
Endothelial Cell Density | baseline, 1 month, 3 months and 6 months after surgery
  Measure by Specular Microscope
Vault measured by anterior segment OCT | 2 hours, 1 day, 1 week, 1 month, 3 months and 6 months after surgery
  Vault measured by anterior segment OCT
Intraocular Pressure | baseline, 1 day, 1 week, 1 month, 3 months and 6 months after surgery
  Intraocular Pressure measured by non-contact tonometers
Refractive error (by Phoropter) | baseline, 1 day, 1 week, 1 month, 3 months and 6 months after surgery
  subjective refraction by Phoropter
Anterior chamber reaction (by a laser flare meter) | baseline, 2 hours, 1 day, 1 week after surgery
  anterior chamber flare value was examined by a laser flare meter
Duration of operation | at the time of the surgery
  Time from the first incision is made to the end of the surgery
Complications of ICL implantation | up to 6 months after surgery
  Lens opacities, Cataract surgery, Pupillary block, Ocular hypertension or glaucoma

CONTACTS AND LOCATIONS:
Overall Officials: AYong Yu, MD. PhD., Principal Investigator — Wenzhou Medical University
Locations (5):
- China (5):
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - The Eye Hispital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Peking Union Medical College Hospital, Beijing
  - Shanghai Ninth People's Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No